CLINICAL TRIAL: NCT02365610
Title: A Double Blind, Randomized, Placebo-controlled, Two-part Study to Investigate the Pharmacokinetics, Followed by Efficacy and Safety of GWP42006 as add-on Therapy in Patients With Inadequately Controlled Focal Seizures.
Brief Title: A Study of GWP42006 in People With Focal Seizures - Part B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWEP1330 Part B; 2014-002594-11 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-19 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy; Focal Seizures
Keywords: Cannabidivarin; CBDV; GWP42006
MeSH Terms: conditions — Epilepsy; Seizures | interventions — cannabidivarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GWP42006 (Experimental): GWP42006
  Interventions: Drug: GWP42006
- Placebo control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: GWP42006
  Other Names: Cannabidivarin; CBDV
  Arms: GWP42006
Drug: Placebo Control
  Other Names: Placebo
  Arms: Placebo control

SUMMARY:
To investigate the potential antiepileptic effects of GWP42006 as add-on therapy in subjects with inadequately controlled focal seizures.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo controlled, two-part study. Part B only will be described in this record.

Subjects who satisfy all inclusion and none of the exclusion criteria will enter a four-week baseline period, followed by a two-week dose escalation period (400 mg twice daily for one week, then 600 mg twice daily for one week), a six-week stable treatment period (800 mg twice daily) and a 12-day taper period. Subjects will be required to attend eight study visits. A follow-up phone call will take place four weeks after last dose.

Subjects will be randomized to receive in a 1:1 ratio, GWP42006 or placebo. Subjects will be required to record a daily diary with information about their seizures, investigational medicinal product (IMP) and concomitant antiepileptic drug (AED) administration.

ELIGIBILITY:
For inclusion in Part B of the study patients must fulfil ALL of the following criteria:

* Male or female aged between 18 and 65 years, inclusive.
* Well-documented history of focal epilepsy, compatible electroencephalogram and clinical history.
* Documented computerized tomography / magnetic resonance imaging that shows no progressive neurologic abnormality.
* Has focal seizures despite prior treatment with at least two AEDs (whether as monotherapies or in combination).
* Currently treated with one to three AEDs.
* All medications or interventions for epilepsy (including ketogenic diet) must have been stable for one month prior to screening and the subject is willing to maintain a stable regimen throughout the study.
* Subject is willing to keep any factors expected to affect seizures stable (such as the level of alcohol consumption and smoking).

The patient may not enter Part B of the study if ANY of the following apply:

* Time of onset of focal epilepsy treatment is less than two years prior to enrolment.
* Patient has seizures that are not of focal onset.
* Patient only has focal seizures without impairment of consciousness or awareness and without an observable motor component (even if autonomic component is present).
* Episode(s) of status epilepticus during one year prior to screening.
* History of pseudo-seizures.
* Vagus Nerve Stimulation, Deep Brain Stimulation, Responsive Neurostimulator System or other epilepsy neurostimulation device have been implanted or activated less than one year prior to screening, and/or stimulation parameters have been stable for less than one month, and/or battery life of unit not anticipated to extend for duration of trial.
* Had epilepsy surgery within one year of screening.
* Subject has clinically significant unstable medical conditions other than epilepsy.
* Subject has an illness in the four weeks prior to screening or randomization, other than epilepsy, which in the opinion of the investigator would affect seizure frequency.
* Subject has significantly impaired hepatic function at Visit 1.
* Active suicidal plan/intent in the past six months, or a history of suicide attempt in the last two years, or more than one lifetime suicide attempt .
* Subject is currently using or has in the past used recreational or medicinal cannabis, or cannabinoid based medications within the three months prior to screening and is unwilling to abstain for the duration for the study.
* Subject has taken St John's Wort in the last two weeks and/or is unwilling to abstain throughout the study.
* Subject has consumed grapefruit or grapefruit juice three days prior to randomization and/or unwilling to abstain in the three days prior to Visits B2 and B7.
* Any known or suspected hypersensitivity to cannabinoids, sesame oil or any of the excipients of the IMP(s).
* Subjects who have received an IMP within the 12 weeks prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline to the end of treatment in focal seizure frequency in subjects taking GWP42006 compared to placebo. | Day -28 to Day 57

SECONDARY OUTCOMES:
Number of subjects considered treatment responders. | Day -28 to Day 57
Change from baseline in seizure subtypes frequency. | Day -28 to Day 57
Change from baseline in composite seizure score. | Day -28 to Day 57
Change from baseline in the number of focal seizure free days. | Day -28 to Day 57
Change from baseline in the usage of rescue medication. | Day -28 to Day 57
Subject Global Impression of Change (SGIC). | Day 57
Physician Global Impression of Change (PGIC) at the end of treatment. | Day 57
The incidence of adverse events as a measure of subject safety. | Day -28 to Day 96

CONTACTS AND LOCATIONS:
Locations (26):
- Czechia (4):
  - Havířov
  - Hradec Králové
  - Prague
  - Rychnov nad Kněžnou
- Hungary (6):
  - Budapest
  - Esztergom
  - Hódmezővásárhely
  - Kecskemét
  - Pécs
  - Szombathely
- Italy (3):
  - Bologna
  - Pavia
  - Rome
- Poland (7):
  - Bydgoszcz
  - Elblag
  - Golub-Dobrzyń
  - Katowice
  - Krakow
  - Warsaw
  - Wroclaw
- Spain (2):
  - Barcelona
  - Madrid
- United Kingdom (4):
  - Birmingham
  - Glasgow
  - Great Yarmouth
  - Stoke-on-Trent

REFERENCES:
- [Derived] Brodie MJ, Czapinski P, Pazdera L, Sander JW, Toledo M, Napoles M, Sahebkar F, Schreiber A; GWEP1330 Study Group. A Phase 2 Randomized Controlled Trial of the Efficacy and Safety of Cannabidivarin as Add-on Therapy in Participants with Inadequately Controlled Focal Seizures. Cannabis Cannabinoid Res. 2021 Dec;6(6):528-536. doi: 10.1089/can.2020.0075. Epub 2021 Feb 15. PMID 33998885